CLINICAL TRIAL: NCT01910558
Title: The Effect of Oral Alpha-Cyclodextrin on Fecal Fat Excretion
Acronym: FAT ABSORBER
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Cancelled by Sponsor
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Quest Nutrition LLC (Unknown)
Responsible Party: Principal Investigator, Frank Greenway, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PBRC 2013-043
Record Dates: First submitted 2013-07-22; First posted 2013-07-29 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Obesity; Cardiovascular Disease
Keywords: Alpha-cyclodextrin; Dietary fiber; Fecal fat; Saturated fat
MeSH Terms: conditions — Obesity; Cardiovascular Diseases | interventions — alpha-cyclodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Alpha-cyclodextrin and digestible starch (Active Comparator): Supplementation with three grams alpha cyclodextrin with three grams of digestible starch
  Interventions: Dietary Supplement: Alpha-cyclodextrin
- Alpha-cyclodextrin (Experimental): Supplementation with six grams of alpha-cyclodextrin
  Interventions: Dietary Supplement: Alpha-cyclodextrin and digestible starch
- Digestible Starch (Placebo Comparator): Supplementation with six grams of digestible starch
  Interventions: Dietary Supplement: Digestible starch

INTERVENTIONS:
Dietary Supplement: Alpha-cyclodextrin and digestible starch — Weight maintaining diet (40% fat, 30% protein, and 30% carbohydrate) supplemented with 3 gram alpha-cyclodextrin and 3 gram of starch
  Arms: Alpha-cyclodextrin
Dietary Supplement: Alpha-cyclodextrin — Weight maintaining diet (40% fat, 30% protein, and 30% carbohydrate) supplemented with 6 grams alpha-cyclodextrin
  Arms: Alpha-cyclodextrin and digestible starch
Dietary Supplement: Digestible starch — Weight maintaining diet (40% fat, 30% protein, and 30% carbohydrate) supplemented with 6 grams digestible starch
  Arms: Digestible Starch

SUMMARY:
Saturated fat leading to elevated low density lipoprotein (LDL) cholesterol is considered a cardiovascular risk factor. The properties associated with α- cyclodextrin, allow it to selectively reduce saturated fat and calories which will have a medically beneficial effect on LDL cholesterol and obesity. The purpose of the research is to evaluate this effect of α- cyclodextrin. It is hypothesized that alpha cyclodextrin supplementation will increase fecal fat on a high saturated fat diet compared to the same diet supplemented with a digestible carbohydrate control

DETAILED DESCRIPTION:
Alpha-cyclodextrin which functions as a soluble dietary fiber, has been shown to a form a stable emulsion with dietary fat in the ratio of 1:9, with a higher affinity for saturated fat compared to unsaturated fat. In humans, supplementation with α-cyclodextrin has been shown to lead to a significant weight loss regardless of whether energy intake was maintained or increased.The aim of this study is to evaluate the results of a 72 hour fecal fat test using stool markers on the last three days of each of three six-day feeding periods. Subjects will be served a weight maintaining diet containing 40% fat (of which 40% will be saturated), 30% protein and 30% carbohydrate for 18 days. Subjects will also consume 1 gram alpha cyclodextrin with 1 gram of starch, 2 grams of alpha cyclodextrin, or 2 grams of starch in capsule form before breakfast, lunch, and dinner every day in each of the three six-day feeding periods. At this dose, alpha-cyclodextrin is recognized as safe by the FDA. All stools will be collected over a 72 hour period at the end of each feeding period and analyzed for fecal fat excretion.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 20 and 30 kg/m2 inclusive
* Weight ≥ 65 kg for females, and ≥ 55 kg for males

Exclusion Criteria:

* Pregnant or nursing.
* Diabetes Mellitus
* Any medication to reduce lipids
* History of gastrointestinal surgery, except for cholecystectomy or appendectomy
* History of malabsorption

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Fecal Fat Excretion compared at three time periods. | Assessment of change at each fourth, fifth, and sixth day of each feeding period.
  Each subject will consume a different product every six consecutive days which is called a feeding period. On the fourth, fifth, and sixth day of each feeding period, a comparison of fat excretion will be measured through a stool sample. These feeding periods will occur for three consecutive six days totaling eighteen days of feeding. 6+6+6=18

SECONDARY OUTCOMES:
Adverse events | The duration of the 18 days in the study.
  Subjects will be asked if they experienced any adverse events. All adverse events will be recorded and evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Frank L Greenway, M.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Background] Comerford KB, Artiss JD, Jen KL, Karakas SE. The beneficial effects of alpha-cyclodextrin on blood lipids and weight loss in healthy humans. Obesity (Silver Spring). 2011 Jun;19(6):1200-4. doi: 10.1038/oby.2010.280. Epub 2010 Dec 2. PMID 21127475
- [Background] Grunberger G, Jen KL, Artiss JD. The benefits of early intervention in obese diabetic patients with FBCx: a new dietary fibre. Diabetes Metab Res Rev. 2007 Jan;23(1):56-62. doi: 10.1002/dmrr.687. PMID 17013969
- [Background] Artiss JD, Brogan K, Brucal M, Moghaddam M, Jen KL. The effects of a new soluble dietary fiber on weight gain and selected blood parameters in rats. Metabolism. 2006 Feb;55(2):195-202. doi: 10.1016/j.metabol.2005.08.012. PMID 16423626